CLINICAL TRIAL: NCT05721261
Title: Regeneration of Acutely Injured Nerves With Temporary Electrical Stimulation
Acronym: REGAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Epineuron Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EPNR-CIP-002
Record Dates: First submitted 2023-02-01; First posted 2023-02-09 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Nerve Injury

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active treatment (Experimental)
  Interventions: Device: Temporary Peripheral Nerve Stimulation System
- Sham treatment (Sham Comparator)
  Interventions: Device: Sham Temporary Peripheral Nerve Stimulation System

INTERVENTIONS:
Device: Temporary Peripheral Nerve Stimulation System — Single use medical device. Therapy consists of single, 1 hour dose of electrical stimulation delivered proximal to injury site.
  Arms: Active treatment
Device: Sham Temporary Peripheral Nerve Stimulation System — Single use medical device. Sham treatment consists of single, 1 hour dose of sham stimulation.
  Arms: Sham treatment

SUMMARY:
A novel temporary peripheral nerve stimulation system that delivers a single dose of electrical stimulation therapy for 1 hour will be evaluated for safety and effectiveness.

ELIGIBILITY:
Inclusion criteria:

* Peripheral nerve injury

Exclusion criteria:

* Peripheral neuropathy
* Patients with any active implanted device

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-08-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Sensory recovery | 6 months
Cumulative incidence of adverse events | 6 months

CONTACTS AND LOCATIONS:
Locations (12):
- United States (5):
  - University of Florida Health, Gainesville, Florida
  - Orlando Health Jewett Orthopedic Institute, Orlando, Florida
  - The Curtis National Hand Center, Baltimore, Maryland
  - WellSpan Health, York, Pennsylvania
  - John Peter Smith Hospital, Fort Worth, Texas
- Canada (7):
  - University of Alberta Hospital, Edmonton, Alberta
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Hamilton General Hospital, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Roth | McFarlane Hand & Upper Limb Centre, London, Ontario
  - North York General Hospital, Toronto, Ontario
  - Trillium Health Partners, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No